CLINICAL TRIAL: NCT04073810
Title: Residual Inflammation and Plaque Progression Long-term Evaluation
Acronym: RIPPLE
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Jason Tarkin, Wellcome Clinical Research Career Development Fellow & Clinical Lecturer, University of Cambridge
Other Study IDs: A095007 (RIPPLE)
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atherosclerosis; Myocardial Infarction; Coronary Artery Disease; Inflammation
MeSH Terms: conditions — Atherosclerosis; Myocardial Infarction; Coronary Artery Disease; Inflammation | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myocardial infarction: Patients with recent MI
  Interventions: Diagnostic Test: PET imaging; Diagnostic Test: Coronary CT angiography; Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: PET imaging — Coronary 68Ga-DOTATATE PET-MRI or PET-CT at baseline and 3 months
Diagnostic Test: Coronary CT angiography — CTCA at baseline and 2 years
Diagnostic Test: Cardiac MRI — Cardiac MRI at 1 year

SUMMARY:
Inflammation drives atherosclerotic plaque rupture triggering most acute coronary syndromes. Despite advances in diagnosis and management of atherosclerosis, patients with myocardial infarction (MI) remain at increased risk of recurrent events. The RIPPLE study aims to examine the relationship between residual coronary inflammation detected by 68Ga-DOTATATE PET in patients treated for MI to long-term plaque progression measured by CT coronary angiography (CTCA). The association between infarct-related myocardial 68Ga-DOTATATE PET and myocardial function and viability will also be assessed.

DETAILED DESCRIPTION:
While vascular inflammation can be detected using 18F-FDG PET, this method lacks inflammatory cell specificity and is unreliable for coronary imaging because of high background signals from the myocardium. Upregulation of somatostatin receptor subtype-2 (SST2) occurs in activated macrophages, offering a novel inflammation imaging target. 68Ga-DOTATATE, an SST2 PET tracer with low myocardial binding, shows promise for imaging coronary inflammation. Having previously demonstrated increased 68Ga-DOTATATE signals in coronary atherosclerotic lesions post-MI, we now aim to study the natural history of residual arterial inflammation in non-culprit arteries and better understand how 68Ga-DOTATATE signals relate to plaque morphology, progression and rupture. Residual infarct-related myocardial inflammation and its association with ischemic myocardial remodelling will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants >18 years old
* Able to give written, informed consent and to lie flat
* First-presentation of myocardial infarction within ~2 weeks
* At least mild non-culprit coronary artery disease on angiography, managed medically

Exclusion Criteria:

* Women of child bearing potential not using adequate contraception
* Contrast allergy or contrast-nephropathy
* Uncontrolled atrial fibrillation
* Chronic kidney disease (eGFR <30 mL/min/1.73 m2)
* Any medical condition, in the opinion of the investigator, that prevents the participant from lying flat during scanning, or from participating in the study
* Uncontrolled chronic inflammatory disorder
* History of recent malignancy deemed relevant to the study by the investigator
* Current use of systemic corticosteroids
* Previous coronary artery bypass grafting surgery (CABG) or percutaneous coronary intervention (PCI) before the index event
* Contraindication to coronary angiography
* Requires CABG or staged non-culprit artery PCI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recent myocardial infarction and medically managed non-culprit coronary artery disease
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
68Ga-DOTATATE PET vs. plaque progression | 2 years
  Comparison of non-culprit coronary artery 68Ga-DOTATATE tissue-to-blood ratio at 12 weeks post-MI in patients with plaque progression (changes in low attenuation plaque volume and total atheroma volume) after 2 years measured by CTCA versus those without

SECONDARY OUTCOMES:
68Ga-DOTATATE PET vs. CTCA-defined plaque morphology | 2 years
  Comparison of coronary 68Ga-DOTATATE imaging to changes in plaque morphology measured by CTCA
68Ga-DOTATATE PET vs. intravascular imaging | Baseline
  Comparison of 68Ga-DOTATATE imaging to plaque morphology defined by high-resolution intravascular imaging performed during invasive coronary angiography
68Ga-DOTATATE PET vs. hsCRP | 2 years
  Comparison of 68Ga-DOTATATE PET to high-sensitivity C-reactive protein
68Ga-DOTATATE PET vs left ventricular myocardial function | 1 year
  Comparison of myocardial 68Ga-DOTATATE PET to left ventricular size and function
68Ga-DOTATATE PET vs myocardial tissue characterization | 1 year
  Comparison of myocardial 68Ga-DOTATATE PET to myocardial scarring and oedema

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Tarkin, MBBS PhD, Principal Investigator — University of Cambridge
Locations (1):
- University of Cambridge, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarkin JM, Joshi FR, Evans NR, Chowdhury MM, Figg NL, Shah AV, Starks LT, Martin-Garrido A, Manavaki R, Yu E, Kuc RE, Grassi L, Kreuzhuber R, Kostadima MA, Frontini M, Kirkpatrick PJ, Coughlin PA, Gopalan D, Fryer TD, Buscombe JR, Groves AM, Ouwehand WH, Bennett MR, Warburton EA, Davenport AP, Rudd JH. Detection of Atherosclerotic Inflammation by 68Ga-DOTATATE PET Compared to [18F]FDG PET Imaging. J Am Coll Cardiol. 2017 Apr 11;69(14):1774-1791. doi: 10.1016/j.jacc.2017.01.060. PMID 28385306
- [Background] Pedersen SF, Sandholt BV, Keller SH, Hansen AE, Clemmensen AE, Sillesen H, Hojgaard L, Ripa RS, Kjaer A. 64Cu-DOTATATE PET/MRI for Detection of Activated Macrophages in Carotid Atherosclerotic Plaques: Studies in Patients Undergoing Endarterectomy. Arterioscler Thromb Vasc Biol. 2015 Jul;35(7):1696-703. doi: 10.1161/ATVBAHA.114.305067. Epub 2015 May 14. PMID 25977567
- [Background] Rominger A, Saam T, Vogl E, Ubleis C, la Fougere C, Forster S, Haug A, Cumming P, Reiser MF, Nikolaou K, Bartenstein P, Hacker M. In vivo imaging of macrophage activity in the coronary arteries using 68Ga-DOTATATE PET/CT: correlation with coronary calcium burden and risk factors. J Nucl Med. 2010 Feb;51(2):193-7. doi: 10.2967/jnumed.109.070672. Epub 2010 Jan 15. PMID 20080898
- [Derived] Corovic A, Wall C, Nus M, Gopalan D, Huang Y, Imaz M, Zulcinski M, Peverelli M, Uryga A, Lambert J, Bressan D, Maughan RT, Pericleous C, Dubash S, Jordan N, Jayne DR, Hoole SP, Calvert PA, Dean AF, Rassl D, Barwick T, Iles M, Frontini M, Hannon G, Manavaki R, Fryer TD, Aloj L, Graves MJ, Gilbert FJ, Dweck MR, Newby DE, Fayad ZA, Reynolds G, Morgan AW, Aboagye EO, Davenport AP, Jorgensen HF, Mallat Z, Bennett MR, Peters JE, Rudd JHF, Mason JC, Tarkin JM. Somatostatin Receptor PET/MR Imaging of Inflammation in Patients With Large Vessel Vasculitis and Atherosclerosis. J Am Coll Cardiol. 2023 Jan 31;81(4):336-354. doi: 10.1016/j.jacc.2022.10.034. PMID 36697134